CLINICAL TRIAL: NCT05327647
Title: A Phase II Randomized Trial of Bicalutamide in Patients Receiving Intravesical BCG for Non-muscle Invasive Bladder Cancer
Brief Title: A Phase II Trial of Bicalutamide in Patients Receiving Intravesical BCG for Non-muscle Invasive Bladder Cancer
Acronym: BicaBCa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Cancer Research Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: MP-20-2022-6318
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non-Muscle Invasive Bladder Cancer
Keywords: Bicalutamide; BCG instillation; Placebo
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — bicalutamide; Nonsteroidal Anti-Androgens

STUDY DESIGN:
Intervention Model Description: The study started with cohort A (open-label study) for around 40 participants. Then the recruitment in cohort A will stop and the recruitment in cohort B (double-blind, with placebo) will start.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bicalutamide (Experimental): Induction intravesical Bacille Calmette-Guérin treatment with 150 mg daily oral bicalutamide for 90 days (in cohort A and cohort B)
  Interventions: Drug: Bicalutamide
- Control Arm (Active Comparator): cohort A: Induction intravesical Bacille Calmette-Guérin treatment
  cohort B: Induction intravesical Bacille Calmette-Guérin treatment with 150 mg daily oral placebo for 90 days
  Interventions: Biological: Control Arm

INTERVENTIONS:
Drug: Bicalutamide — Induction intravesical BCG with bicalutamide 150 mg for 90 days
  Other Names: Nonsteroidal antiandrogen
  Arms: Bicalutamide
Biological: Control Arm — Induction BCG
  Arms: Control Arm

SUMMARY:
This is a phase II randomized controlled clinical trial comparing standard induction BCG versus bicalutamide and standard induction BCG among patients with non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
Bladder cancer is the second most common urological cancer after prostate cancer. Non-muscle invasive bladder cancer (NIMBC) is the most common form (~ 75%). The standard treatment involves the use of intravesical instillation of bacillus Calmette-Guérin (BCG). Nonetheless, 30-40% of the patients still relapse or progress. Clinical and laboratory research suggests that medications targeting the androgen receptor, such as bicalutamide, combined with the standard treatment with BCG may decrease the recurrence rate of NMIBC.

The study is composed of two cohort A (open-label, around 40 patients) and B (double-blind, with placebo, around 120 patients).

In the cohort A, the participants will be randomized to either the treatment with 1) daily intake of 150 mg bicalutamide for 3 months overlapping with the 6 cycles of intravesical instillations of BCG or 2) the standard of care of 6 cycles of intravesical instillation BCG.

In the cohort B, the participants will be randomized to either the treatment with 1) daily intake of 150 mg bicalutamide for 3 months overlapping with the 6 cycles of intravesical instillations of BCG or 2) daily intake of 150mg placebo for 3 months + the standard of care of 6 cycles of intravesical instillation BCG.

The participation in this trial should last 36 months from the screening visit to the last follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Males, age 18 or greater.
2. Patients with histologically confirmed non-muscle invasive urothelial carcinoma.
3. Patients have been recommended for a course of intravesical BCG induction treatment by their urologist
4. Patients who received gemcitabine, epirubicin or mitomycin C instillations immediately post-operatively will be eligible for enrollment.
5. Patients with partners of child-bearing potential must agree to 2 acceptable forms of birth control and be continued for at least 3 months after study drug is discontinued.

Exclusion Criteria:

1. Patients who have received induction BCG therapy within the last 5 years will be ineligible for enrolment.
2. Patients with a history of myocardial infarction or hospital admission for heart failure within the previous 12 months or who have unstable cardiovascular status will be ineligible for enrolment.
3. Patients who have uncontrolled hypertension (for our purposes, defined as those having a systolic blood pressure > 160 documented on 2 occasions despite appropriate medical therapy) will similarly be ineligible.
4. Patients with a history of liver disease whose hepatic enzymes, alkaline phosphatase or bilirubin are greater than twice the upper limit of normal will be ineligible.
5. Patients with clinical hypogonadism, those on androgen replacement therapy, or those with prostate cancer or other diseases treated with systemic hormonal therapy will be ineligible for study enrolment. Patients receiving 5ARIs will not be excluded.
6. Patients who have cancer treatment ongoing or planned in the near future which can be anticipated to decrease their 2-year survival or BCa treatment plan will be ineligible.
7. Patients taking an investigational drug within 2 weeks of enrolment into this study will be ineligible.
8. Patients receiving or planning to receive coumadin therapy will be ineligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of bladder tumour recurrence | 3 years
  To time to bladder tumor recurrence compared to the standard of care induction BCG

SECONDARY OUTCOMES:
Incidence of tumour progression | 3 years
  To compare the incidence of tumor progression between the intervention and control arms
Number of tumor recurrences | 3 years
  To compare the overall incidence of tumor recurrences between intervention and control arms
Number of tumours at first recurrence | 3 years
  Evaluation of the number of tumours at first recurrence between the two arms
Quality of life (QLQ-C30) | 3 years
  Evaluation of quality of life with QLQ-C30 questionnaire (EORTC Core Quality of Life questionnaire). The scale scores range from 0 to 100. A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptom
Evaluation of urinary symptoms | 3 years
  Evaluation of urinary symptoms with International Prostate Symptom Score (IPSS) . questionnaire. The total score can range from 0 to 35 (0 being asymptomatic and 35 being very symptomatic).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Toren, MD,PhD,FRCSC, Study Chair — CHU de Québec-Université Laval; Wassim Kassouf, MDCM,FRCSC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Melissa Huynh, MD,MPH,FRCSC, Principal Investigator — London Health Sciences Centre, Victoria Hospital; Jean-Baptiste Lattouf, MD,FRCSC, Principal Investigator — Centre Hospitalier Universitaire de Montréal (CHUM); Girish Kulkarni, BSc, MD, PhD, FRCSC, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (7):
- Canada (7):
  - London Health Sciences Centre, London, Ontario
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre intégré de santé et services sociaux de Chaudière Appalaches, Lévis, Quebec
  - Centre Hospitalier de l'Université De Montréal_CHUM, Montreal, Quebec
  - McGill University Health Centre_CUSM, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No